CLINICAL TRIAL: NCT05525897
Title: A Multi-case Feasibility Study for an Introductory Psychoeducational Course (Life Skills 101) for Students in Higher Education
Brief Title: Life Skills 101 Feasibility Study
Acronym: LEVELUP1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cyprus (Other)
Collaborators: VU University of Amsterdam (Other); University of Crete (Other); University of Jaén (Other)
Responsible Party: Principal Investigator, Prof. Georgia Panayiotou, Dr. Georgia Panayiotou, Professor of Clinical Psychology, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LEVELUP_Feasibility1
Record Dates: First submitted 2022-08-12; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Soft Skills
Keywords: Soft skills; transversal skills; life skills; 21st century skills

STUDY DESIGN:
Intervention Model Description: The investigators will use a pre-post design with a multi-case study approach to evaluate the feasibility and implementation of the psycho-educational intervention in four university settings.
  In specific, three universities (CY, GR, SP) will run a single-arm study, while the fourth university (NL) will run an RCT pilot study (see RCT pilot study methods for details).
  A mixed-methods design will be used to determine the feasibility and acceptability of a novel soft-skills psychoeducational course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life skills course (Experimental): Participants will take part in the psychoeducational course
  Interventions: Other: Psychoeducational
- Waitlist (No Intervention)

INTERVENTIONS:
Other: Psychoeducational — The focus of the course is to teach students the fundamental theories, and practices of soft skills, as well as providing cases and material that give students the opportunity to learn from real life experiences.
  Arms: Life skills course

SUMMARY:
In the present study, the investigators aim to examine the feasibility of embedding a classroom-based soft skills intervention within a tertiary curriculum.

The primary objective of this study is to assess the acceptability and feasibility of the "Life Skills 101", a novel psychoeducational course for students in higher education.

The secondary objective of this study is to evaluate potential effectiveness of the course by measuring students' acquired knowledge and improvement on self-insight.

Different methodologies will be used as part of the stage model for behavioral intervention development. In specific, three universities (CY, GR, SP) will run a single-arm study, while the fourth university (NL) will run an RCT pilot study.

DETAILED DESCRIPTION:
Background/Rationale The role of Higher Education in sustained economic growth, and social progress is critical. HE institutions (HEIs) as key 'future shaper' settings, host a significant proportion of talented youth, future workforce, and leaders. Entering university marks a turning point for youth, since HEIs can empower young people to transform and expand skills to manage complex and global environmental and societal challenges.

Soft skills, such as the ability to set goals and achieve them, to regulate emotions, to demonstrate agility and adaptability, and manage interpersonal relationships, are now an emerging trend for tackling global economic and societal challenges. Despite soft skills importance, evidence confirms a "skills gap", meaning that youth lack soft skills that are highly important in the workplace. In addition, soft skills related to mental and physical health, wellbeing and adjustment, have received growing interest over recent years, and have become even more critical in the context of emerging needs to build resilience in the face of the Covid-19 pandemic and in preparation for future crises.

Given these challenges to individuals' academic performance, work achievement, mental health, it would be advisable to equip students with the resources required for life success. As these skills become increasingly of central interest to communities, it becomes a pertinent question on how to expand them within the academic context by learning relevant information and practicing skills in a way that is responsive to the needs of the wider student community. A key priority for HEIs is to promote a comprehensive approach to education, by putting students' transversal skills on an equal footing with profession-specific knowledge and skills. One efficient way to address this, in a way that can reach as many interested students as possible, is through incorporating the necessary material in existing, popular and frequently offered elective or mandatory courses, in which training these skills is suitable.

In the present study, the investigators aim to examine the feasibility of embedding a classroom-based soft skills intervention within a tertiary curriculum. This course covers cutting-edge research on how people acquire self-regulatory skills enabling them to achieve personal, academic, and professional goals. Students will learn through instruction and experiential methods, how these discoveries relate to needs, cognitions, emotions, and behaviors, and what tools can be used to achieve their goals.

Study aims/Objectives

The primary objective of this study is to assess the acceptability and feasibility of the "Life Skills 101", a novel psychoeducational course for students in higher education. The secondary objective of this study is to evaluate potential effectiveness of the course by measuring students' acquired knowledge and improvement on self-insight. The specific objectives of the study are to:

1. Determine feasibility and acceptability of the psychoeducational soft skills intervention.

   1. To estimate feasible recruitment and refusal rates.
   2. To measure key outcome domains such as completion rates, missing data, students-reported measures of social satisfaction.
   3. To determine the acceptability of course resources and factors influencing this.
   4. To measure participants' willingness to participate in highly specialized soft skills training.
2. Estimate effectiveness in terms of changes over time in knowledge, improvement in self-insight and psychological flexibility.
3. Use findings to refine the program and inform the development of a future large-scale randomised control trial (RCT).
4. Explore associated changes in mental health (only RCT pilot).

ELIGIBILITY:
Inclusion Criteria

- People who are enrolled as students in one of the four universities.

Exclusion criteria

- No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability | up to 10 weeks
  At post-intervention, all participants will complete a course satisfaction/acceptability questionnaire. The questionnaire will consist of two parts: In part A (quantitative) students will be asked several Likert-scale questions, while part B (qualitative) while contain open-ended response questions relating to their experience, satisfaction, and the challenges/enablers associated with design and implementation of the course.
  Qualitative data from open-ended questions will be considered alongside the quantitative measures to assess the feasibility of the intervention. The feasibility and acceptability of the intervention will be evaluated, using multiple primary endpoints such as:
  1. Adherence (Total registrations, Attendance Rates, Homework Adherence, Dropouts, App Downloads, App use)
  2. Acceptability (Course acceptability, course satisfaction, perceptions measured by both Likert Scale Questionnaire and open-ended questions).
Self-efficacy | up to 10 weeks
  The General self-efficacy scale (GSE) consists of 10-items on a 4-point Likert scale (1 'not at all true' to 4 'exactly true'). A total score, on a scale of 10 to 40 can be calculated. Higher scores indicate higher perceived general self-efficacy. Its internal consistency is good (Cronbach α = .85).

SECONDARY OUTCOMES:
Knowledge | up to 10 weeks
  The research team will develop a 10-item multiple choice quiz to assess students' knowledge on fundamental concepts of the course content.
Self-Reflection and Insight Scale- Short Form | up to 10 weeks
  Self-Reflection and Insight Scale- Short Form (SRIS-SF) to assess students' changes in the clarity of understanding their thoughts, feelings and behavior (Self-Reflection Cronbach's α = .87 and Insight Scale Cronbach's α = .83). Higher total score mean more perceived levels of self-awareness.
Private Self-Consciousness (PrSC) dimension of Self-Consciousness Scale | up to 10 weeks
  Private Self-Consciousness (PrSC) dimension of Self-Consciousness Scale (SCS; Cronbach's α = .79), measures internal state awareness, the tendency to cover aspects of self, such as values, beliefs, feelings etc. Higher score refers to higher levels of self-consciousness.
Single-item self-assessment questions | up to 10 weeks
  Single-item self-assessment questions (about students' perceived competency on the skill taught) will be filled (pre-post session) via a digital learning tool (app). The question will be posed as follows: "Imagine a ladder (see picture), which represents how competent a person is according to a skill. The top of the ladder reflects the mastery of skill, while the bottom reflects significant deficiencies in that skill. At what point on the ladder would you place yourself in Self-regulation skills? Choose the number that best represents you where you place yourself: 1-10".
Psychological flexibility | up to 10 weeks
  The Acceptance and Action Questionnaire-II is a 7-item measure of psychological flexibility rated on a 7-point scale (Cronbach's α = 0.84). It assesses the ability to be fully present in the moment and adjusting behaviors based on the situational demands, personal values and goals. Higher total score mean less flexibility.
Positive mental health | up to 10 weeks
  Mental health Continuum-Short Form (MHC-SF) consists of 14-items on a 6- point Likert scale (0 'never' to 5 'everyday'). It measures (1) emotional wellbeing (happiness, interest, satisfaction); (2) psychological wellbeing (self-acceptance, mastery, positive relations, personal growth, autonomy, purpose in life), and (3) social wellbeing (social contribution, integration, actualization, acceptance, coherence). Higher scores indicate greater levels of positive well-being. The instrument has shown good internal reliability for the total score (Cronbach's α = .89) and acceptable to good internal consistency for its subscales (Cronbach's α = .74 to 83).
Depression, anxiety and stress | up to 10 weeks
  Depression Anxiety Stress Scales (DASS-21) consist of three scales (7 items per scale) measuring states of depression, anxiety and stress on a 4 point Likert scale (0 'almost always' to 4 'never'). higher scores indicating a greater number of symptoms. The DASS-21 subscales show good internal consistency (Cronbach's α = 0.81- 0.88).
Trait worry | up to 10 weeks
  Penn state Worry Questionnaire (PSWQ) is a self-report questionnaire measuring frequent negative thoughts. The scale has 14 items and have to be scored on a 4 point scale with 0=not true and 4=very true. Higher scores are indicative of higher levels of trait worry. The instrument shows excellent internal consistency (Cronbach α = .91).
Personal growth mindset | up to 10 weeks
  The Personal Growth Initiative Scale - II © (PGIS-II) measures the active and intentional involvement in personal change and development in terms of readiness to change, planfulness, using resources, and intentional behavior. Higher scores are indicative of greater Personal Growth Initiative. The instrument's internal consistency is excellent (Cronbach's α = .90 to .94).

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Panayiotou, PhD, Principal Investigator — University of Cyprus
Locations (4):
- University of Cyprus, Nicosia, Cyprus
- University of Crete, Rethymno, Greece
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands
- Universidad de Jaén, Jaén, Spain

IPD SHARING:
Plan to Share IPD: Undecided